CLINICAL TRIAL: NCT04275700
Title: Study of Ovarian Function Following Intraovarian Injection of Platelet Rich Plasma (PRP) In Women With Evidence of Diminished Ovarian Function
Brief Title: Study of PRP in Women With Evidence of Diminished Ovarian Reserve
Acronym: PRP4AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Human Reproduction (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09182018-01
Record Dates: First submitted 2018-10-22; First posted 2020-02-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Diminished Ovarian Reserve; Ovarian Failure
Keywords: Platelet Rich Plasma

STUDY DESIGN:
Intervention Model Description: Each Ovary will be injected with A-PRP.
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A-PRP (Experimental): The cortex of each ovary will be injected with autologous platelet rich plasma.
  Interventions: Procedure: A-PRP

INTERVENTIONS:
Procedure: A-PRP — The cortex of each ovary will be injected with autologous platelet rich plasma. Up to seven different sites will be injected under ultrasound guidance. The patient will be under IV sedation.
  Other Names: Autologous Platelet Rich Plasma

SUMMARY:
The hypothesis of the study is that ovaries of women with a history of poor response to ovulation induction may benefit from exposure to growth factors known to be present in Platelet Rich Plasma (PRP). Since even ovaries from women with poor response still contain primordial follicles (which, however, no longer undergo recruitment), it is hoped that PRP injections into ovaries will activate follicular recruitment pathways and, subsequently, result in follicle growth. Should such growth be observed, follicles will be supported with routine daily gonadotropin stimulation until hCG trigger.

DETAILED DESCRIPTION:
The hypothesis of the study is that ovaries of women with a history of poor response to ovulation induction may benefit from exposure to growth factors known to be present in PRP.

Autologous Platelet Rich Plasma (A-PRP) is plasma with a concentration of platelets above the blood baseline. A-PRP is developed from autologous blood. Within A-PRP, the concentration of platelets delivers an increased number of growth factors. In this study A-PRP will be prepared using Regen Lab PRP Kit which is approved by US-FDA for preparation of PRP.

PRP is becoming widely used in a variety of medical procedures seeking tissue remodeling and/or healing as an intervention. To date, applications in orthopedics, wound healing, dermatology and plastic surgery have gained general acceptance, primarily as the role of platelets and their activation in tissue repair and recovery has become better understood at a cellular and molecular level. This knowledge base provides a foundation for the present study because of the ready availability of FDA-approved kits for autologous PRP preparations and the recognition that the aging ovary acquires tissue pathologies in the form of wound healing and fibrosis as a result of repeat ovulations over the reproductive lifespan of women. Since PRP is an autologous blood product, and is widely used via injection into various organs and tissues, safety concerns are minimal.

This study will involve only adult women with a diagnosis of diminished ovarian reserve. All consenting participants will receive injections of autologous Platelet RIch Plasma (A-PRP) in both ovaries under ultrasound guidance performed after induction of IV sedation.

Assumption of this study is that in women with previous poor response to ovulation induction will show limited follicle growth. The study will try to estimate effect of PRP on this condition by comparing post-PRP response to the previous response. The investigators recognize that there will be a possibility of apparent response based on regression to the mean. The investigators expect that study of fifty patients should be enough to determine if there is a potential clinical effect and to allow estimation of that effect for power calculations for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Women with failure to respond well to ovulation induction by having fewer than 1 cleavage stage embryo in response to past ovulation induction who do not qualify for the PRP4POI study
* Age 54 years and under.
* FSH > 12
* AMH < 1.1
* -No Aspirin or Motrin for one week before treatment

Exclusion Criteria:

* Age > 54 years
* Marked thrombocytopenia
* Blood diseases
* Hypofibrinogenemia
* Hemodynamic instability
* Anticoagulant or antiaggregant treatment
* Oncological diseases (specially, skeletal system and blood)
* Sepsis
* Acute and chronic infectious diseases
* Autoimmune diseases, for example, lupus erythematosus, etc.

Relative contraindications for PRP

* Chronic liver diseases in the exacerbation phase
* Chronic intoxication against the background of long-term use of alcohol, addictive drugs, an administration of potent medications
* Use of steroidal anti-inflammatory drugs in less than 2 days before drawing the blood, an injection of corticosteroids in little less than 2 weeks before the procedure
* Pregnancy
* Inflammatory skin diseases, chronic dermatosis in the exacerbation phase, for example, psoriasis, atopic eczema, etc.

Ages: 21 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Emergence of new ovarian follicles with evidence of estradiol production | Change from baseline to 12 weeks
  Emergence of new ovarian follicles greater than 4 mm in average diameter as measured using pelvic sonography with evidence of change estradiol serum estradiol levels as measured using a immuno assay.

SECONDARY OUTCOMES:
Change in serum AMH | Change from baseline to 12 weeks
  Increase in serum AMH from baseline level as measured using an immuno assay
Number of participants with retrieval of oocytes in an IVF cycle | 6 months
  Number of participants with retrieval of oocytes in an IVF cycle
Number of participants that establish a Clinical Pregnancy | 12 months
  Number of participants that establish a Clinical Pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Gleicher, MD, Study Chair — Medical Director
Locations (1):
- Center For Human Reproduction, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual patient data.

REFERENCES:
- [Background] Barad DH, Albertini DF, Molinari E, Gleicher N. Preliminary report of intraovarian injections of autologous platelet-rich plasma (PRP) in extremely poor prognosis patients with only oocyte donation as alternative: a prospective cohort study. Hum Reprod Open. 2022 Jun 28;2022(3):hoac027. doi: 10.1093/hropen/hoac027. eCollection 2022. PMID 35795849

DOCUMENTS (1):
  • Informed Consent Form (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT04275700/ICF_000.pdf